CLINICAL TRIAL: NCT03663166
Title: Radiation and Chemotherapy With Ipilimumab Followed by Nivolumab for Patients With Stage III Unresectable NSCLC
Brief Title: Radiation and Chemotherapy With Ipilimumab Followed by Nivolumab for Patients With Stage III Unresectable Non-Small Cell Lung Cancer (NSCLC)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Increased SAE occurrence per PI
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MCC-19704
Record Dates: First submitted 2018-09-06; First posted 2018-09-10 (Actual); Results first posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Lung; Unresectable NSCLC; Radiation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Platinum Compounds; Ipilimumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Radiation and Chemotherapy (Experimental): Thoracic Radiotherapy with cytotoxic platinum based chemotherapy with cytotoxic platinum based chemotherapy including cisplatin and etoposide, carboplatin and paclitaxel or cisplatin and pemetrexed (for patients with non-squamous histology) and Ipilimumab.
  Interventions: Radiation: Thoracic Radiotherapy; Drug: Platinum Based Chemotherapy; Drug: ipilimumab
- Nivolumab (Experimental): Nivolumab 480 mg (30 minute IV infusion) after completion of radiation and chemotherapy for up to 12 cycles until progression.
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Radiation: Thoracic Radiotherapy — 2 Gy in 30 fractions directed at all sites of suspected disease
  Arms: Radiation and Chemotherapy
Drug: Platinum Based Chemotherapy — Platinum based chemotherapy including cisplatin and etoposide, carboplatin and paclitaxel or cisplatin and pemetrexed (for patients with non-squamous histology).
  Arms: Radiation and Chemotherapy
Drug: ipilimumab — ipilimumab 1mg/kg delivered concurrently with initiation of chemoradiotherapy and in week 4 of chemoradiotherapy
  Arms: Radiation and Chemotherapy
Drug: Nivolumab — Nivolumab 480 mg (30 minute IV infusion) at least 7 days but no more than 21 days after completion of radiation and chemotherapy every 4 weeks for up to 12 cycles.
  Arms: Nivolumab

SUMMARY:
This study is to determine if Stage III NSCLC patients treated with ipilimumab with thoracic radiation therapy followed by nivolumab monotherapy every 4 weeks for up to 12 months show an improved 12-month Progression Free Survival (PFS) rate compared with a 12-month historical PFS rate of 49% among patients treated in a similar fashion with concurrent chemoradiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Participants must have signed and dated a written informed consent form.
* Participants must be willing and able to comply with proposed visit and treatment schedule.
* Patients with NSCLC documented by histology or cytology from brushing, washing, or needle aspiration of a defined lesion, but not from sputum cytology alone.
* Patients must have presented at initial diagnosis with Stage III disease according to American Joint Committee on Cancer (AJCC) Staging Manual, 8th Edition;
* Patients must be deemed by the treating investigator to be surgically unresectable. I
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 or 1
* Patients must initiate study treatment 60 days from the date of pathologic diagnosis.
* Tumor biopsy specimen including at least formalin-fixed, paraffin-embedded (FFPE) tumor tissue block or 10 unstained slides of tumor sample (archival or recent) for biomarker evaluation must be available for submission to the central lab for correlative studies.
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test within 14 days prior to the start of thoracic radiation therapy.
* Male participants must be willing to refrain from sperm donation during the entire study and for 5 half-lives of study drug plus 90 days (duration of sperm turnover).
* Investigators shall counsel WOCBP and male participants who are sexually active with WOCBP on the importance of pregnancy prevention and the implications of an unexpected pregnancy. Investigators shall advise on the use of highly effective methods of contraception which have a failure rate of </= 1% when used consistently and correctly. Azoospermic males are exempt from contraceptive requirements.
* WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug(s) plus 5 half-lives of study drug (half-life up to 25 days) plus 30 days (duration of ovulatory cycle) for a total of 5 months post-treatment completion.
* WOCBP who are continuously not heterosexually active are exempt from contraception requirements. However, they must still undergo pregnancy testing as described in this section.
* Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug (s) plus 5 half-lives of the study drug (half-life up to 25 days) plus 90 days (duration of sperm turnover) for a total of 7 months post-treatment completion

Exclusion Criteria:

* All toxicities attributed to prior anti-cancer therapy must have been resolved to Grade 1 (NCI CTCAE Version 4) or baseline before administration of study drug(s). Exceptions may apply.
* Women who are pregnant or breastfeeding
* Active, known, or suspected autoimmune disease. Patients with an autoimmune paraneoplastic syndrome requiring concurrent immunosuppressive treatment are excluded. Patients with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll
* A condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of study initiation. Corticosteroids with minimal systemic absorption (inhaled or topical steroids) and adrenal replacement steroid doses > 10 mg daily prednisone equivalent are permitted in the absence of active autoimmune disease
* Prior therapy with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody
* Interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity.
* Any patient requiring supplemental oxygen therapy.
* Previous malignancies (except non-melanoma skin cancers, and some in situ cancers) unless a complete remission was achieved at least 2 years prior to study entry AND no additional therapy is required during the study period.
* Known medical condition that, in the investigator's opinion, would increase the risk associated with study participation or study drug(s) administration or interfere with the interpretation of safety results
* Major surgery or significant traumatic injury that is not recovered at least 14 days before the initiation of thoracic radiation therapy.
* Positive test for hepatitis B virus (HBV) using HBV surface antigen (HBVsAg) test or positive test for hepatitis C virus (HCV) using HCV ribonucleic acid (RNA) or HCV antibody test indicating acute or chronic infection. Individuals with a positive test for HCV antibody but no detection of HCV RNA indicating no current infection are eligible.
* Known medical history of testing positive for human immunodeficiency virus (HIV) or known medical history of acquired immunodeficiency syndrome (AIDS)
* Inadequate hematologic function.
* Inadequate hepatic function.
* Inadequate pancreatic function.
* History of allergy or hypersensitivity to any of the study drugs or study drug components

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2021-10-22 (Actual); Study Completion 2021-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bradford Perez, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (3):
- United States (3):
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - UNC Limeberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina

RESULTS

PARTICIPANT FLOW:
Groups:
- Radiation and Chemotherapy, Followed by Nivolumab: Thoracic Radiotherapy with cytotoxic platinum based chemotherapy with cytotoxic platinum based chemotherapy including cisplatin and etoposide, carboplatin and paclitaxel or cisplatin and pemetrexed (for patients with non-squamous histology) and ipilimumab .
  Thoracic Radiotherapy: 2 Gy in 30 fractions directed at all sites of suspected disease
  Platinum Based Chemotherapy: Platinum based chemotherapy including cisplatin and etoposide, carboplatin and paclitaxel or cisplatin and pemetrexed (for patients with non-squamous histology).
  Ipilimumab: Ipilimumab 1mg/kg delivered concurrently with initiation of chemoradiotherapy and in week 4 of chemoradiotherapy
  Nivolumab 480 mg (30 minute IV infusion) after completion of radiation and chemotherapy for up to 12 cycles until progression.
  Nivolumab: Nivolumab 480 mg (30 minute IV infusion) at least 7 days but no more than 21 days after completion of radiation and chemotherapy every 4 weeks for up to 12 cycles.
Period: Overall Study
Arm/Group | Radiation and Chemotherapy, Followed by Nivolumab
Started | 19
Completed | 18
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Radiation and Chemotherapy, Followed by Nivolumab: Thoracic Radiotherapy with cytotoxic platinum based chemotherapy with cytotoxic platinum based chemotherapy including cisplatin and etoposide, carboplatin and paclitaxel or cisplatin and pemetrexed (for patients with non-squamous histology) and Ipilimumab.
  Thoracic Radiotherapy: 2 Gy in 30 fractions directed at all sites of suspected disease
  Platinum Based Chemotherapy: Platinum based chemotherapy including cisplatin and etoposide, carboplatin and paclitaxel or cisplatin and pemetrexed (for patients with non-squamous histology).
  Ipilimumab: ipilimumab 1mg/kg delivered concurrently with initiation of chemoradiotherapy and in week 4 of chemoradiotherapy
  Nivolumab 480 mg (30 minute IV infusion) after completion of radiation and chemotherapy for up to 12 cycles until progression.
  Nivolumab: Nivolumab 480 mg (30 minute IV infusion) at least 7 days but no more than 21 days after completion of radiation and chemotherapy every 4 weeks for up to 12 cycles.
Arm/Group | Radiation and Chemotherapy, Followed by Nivolumab
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 17
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Unacceptable Toxicity Status at the End of 8-week Safety Observation Period
Description: Unacceptable toxicity defined as:
  * Any grade 4 immune related adverse event (irAE)
  * Any grade 3 irAE, excluding pneumonitis, that does not downgrade to grade 2 within 7 days after onset of the event despite optimal medical management including systemic corticosteroids or does not downgrade to ≤ grade 1 or baseline within 14 days
  * Liver transaminase elevation > 8 × ULN or total bilirubin > 5 × ULN,
  * Any ≥ grade 3 non-irAE, with some exclusions. Result is provided as number of participants with unacceptable toxicity within 8 weeks of commencing study therapy.
Time Frame: At 8 weeks of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation and Chemotherapy, Followed by Nivolumab
Number analyzed (Participants) | 19
Participants | 6

2. Primary Outcome: Percentage of Participants Without Disease Progression at 12 Months
Description: Disease Progression defined as the duration from date of registration to date of first documentation of progression as defined using Response Evaluation Criteria in Solid Tumors (RECIST) v 1.1 and assessed by local investigator or symptomatic deterioration (as defined in Outcome 1) or death due to any cause. Patients last known to be alive without report of progression are censored at date of last disease assessment. For patients with a missing scan (or consecutive missing scans) whose subsequent scan determines progression, the expected date of the first missing scan (as defined by the disease assessment schedule) will be used as the date of progression.
Time Frame: 12 months post treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Radiation and Chemotherapy, Followed by Nivolumab: Thoracic Radiotherapy with cytotoxic platinum based chemotherapy with cytotoxic platinum based chemotherapy including cisplatin and etoposide, carboplatin and paclitaxel or cisplatin and pemetrexed (for patients with non-squamous histology) and Ipilimumab.
  Thoracic Radiotherapy: 2 Gy in 30 fractions directed at all sites of suspected disease
  Platinum Based Chemotherapy: Platinum based chemotherapy including cisplatin and etoposide, carboplatin and paclitaxel or cisplatin and pemetrexed (for patients with non-squamous histology).
  Ipilimumab: Ipilimumab1mg/kg delivered concurrently with initiation of chemoradiotherapy and in week 4 of chemoradiotherapy
  Nivolumab 480 mg (30 minute IV infusion) after completion of radiation and chemotherapy for up to 12 cycles until progression.
  Nivolumab: Nivolumab 480 mg (30 minute IV infusion) at least 7 days but no more than 21 days after completion of radiation and chemotherapy every 4 weeks for up to 12 cycles.
Arm/Group | Radiation and Chemotherapy, Followed by Nivolumab
Number analyzed (Participants) | 19
percentage of participants | 58 [33 to 76]

3. Secondary Outcome: Percentage of Participants Who Experienced 12 Month Distant Metastasis Free Survival (DMFS)
Description: DMFS is defined as the duration from date of registration to date of first documentation of distant metastatic progression beyond the primary tumor site as well as regional lymph nodes assessed by local investigator or symptomatic deterioration (as defined in Outcome 1) or death due to any cause. Patients last known to be alive without report of distant metastatic progression are censored at date of last disease assessment.
Time Frame: 12 months post treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Radiation and Chemotherapy, Followed by Nivolumab
Number analyzed (Participants) | 19
percentage of participants | 63.2 [41.7 to 85]

4. Secondary Outcome: Objective Response Rate (ORR) at 6 Months
Description: ORR is defined as the proportion of all treated subjects whose best overall response is either a complete response or partial response according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria. Best Objective Response (BOR) will also be reported Complete Response (CR) or Partial Response (PR) determinations included in the assessment must be confirmed by a consecutive second (confirmatory) evaluation meeting the criteria for response that is performed at least 4 weeks after the criteria for response are first met. When Stable Disease (SD) is believed to be the best response, it must meet a minimum SD duration of 49 days. Measurements must have met the SD criteria at least once after study entry.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Radiation and Chemotherapy, Followed by Nivolumab
Number analyzed (Participants) | 19
percentage of participants | 66 [41 to 87]

ADVERSE EVENTS:
Time Frame: Adverse Events collected from on study date to 100 days after study drug discontinuation, approximately 14 months.
Arm/Group | Radiation and Chemotherapy, Followed by Nivolumab
All-Cause Mortality (participants affected / at risk) | 9/19
Serious Adverse Events (participants affected / at risk) | 13/19
Other Adverse Events (participants affected / at risk) | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiation and Chemotherapy, Followed by Nivolumab (N=19)
Dehydration (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Lung infection (Infections and infestations) | 3 (6)
Atrial fibrilation (Cardiac disorders) | 2 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (2)
Thromboembolic event (Vascular disorders) | 2 (3)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 (8)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Stroke (Nervous system disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Investigations - Other (Investigations) | 1 (1) — pancytopenia
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiation and Chemotherapy, Followed by Nivolumab (N=19)
Esophagitis (Gastrointestinal disorders) | 13 (19)
Constipation (Gastrointestinal disorders) | 9 (12)
Dysphagia (Gastrointestinal disorders) | 8 (12)
Nausea (Gastrointestinal disorders) | 7 (11)
Diarrhea (Gastrointestinal disorders) | 6 (8)
Vomiting (Gastrointestinal disorders) | 5 (9)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 (4)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 4 (6)
Dry mouth (Gastrointestinal disorders) | 3 (5)
Abdominal pain (Gastrointestinal disorders) | 2 (3)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Hemorrhoids (Gastrointestinal disorders) | 2 (2)
Belching (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 12 (23)
Edema limbs (General disorders) | 5 (6)
Pain (General disorders) | 4 (4)
Chills (Gastrointestinal disorders) | 3 (4)
Fever (General disorders) | 3 (5)
Malaise (General disorders) | 3 (4)
Non-cardiac chest pain (General disorders) | 2 (4)
Flu like symptoms (General disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 10 (22)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (12)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (11)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 5 (7)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Weight loss (Investigations) | 6 (21)
Creatinine increased (Investigations) | 3 (14)
Lipase increased (Investigations) | 3 (8)
Platelet count decreased (Investigations) | 3 (5)
Weight gain (Investigations) | 3 (5)
Alanine aminotransferase increased (Investigations) | 2 (8)
Lymphocyte count decreased (Investigations) | 2 (6)
Neutrophil count decreased (Investigations) | 2 (2)
Serum amylase increased (Investigations) | 2 (5)
White blood cell decreased (Investigations) | 2 (4)
Aspartate aminotransferase increased (Investigations) | 1 (2)
Investigations - Other (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 8 (9)
Dehydration (Metabolism and nutrition disorders) | 6 (8)
Hypokalemia (Metabolism and nutrition disorders) | 4 (6)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (4)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 8 (8)
Insomnia (Psychiatric disorders) | 8 (10)
Confusion (Psychiatric disorders) | 3 (4)
Depression (Psychiatric disorders) | 2 (2)
Agitation (Psychiatric disorders) | 1 (1)
Thrush (Infections and infestations) | 6 (6)
Lung infection (Infections and infestations) | 5 (7)
Sinusitis (Infections and infestations) | 2 (2)
Bronchial infection (Infections and infestations) | 1 (1)
Infections and infestations - Other (Infections and infestations) | 1 (1)
Mucosal infection (Infections and infestations) | 1 (1)
Pelvic infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (4)
Vaginal infection (Infections and infestations) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4 (5)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 4 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 6 (6)
Dysgeusia (Nervous system disorders) | 5 (5)
Headache (Nervous system disorders) | 5 (7)
Stroke (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (2)
Tremor (Nervous system disorders) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 7 (12)
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 2 (3)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1)
Hypotension (Vascular disorders) | 4 (4)
Thromboembolic event (Vascular disorders) | 4 (6)
Hypertension (Vascular disorders) | 3 (4)
Hematoma (Vascular disorders) | 1 (1)
Vascular disorders - Other (Vascular disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 8 (16)
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 2 (3)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 5 (5)
Atrial fibrillation (Cardiac disorders) | 2 (5)
Atrial flutter (Cardiac disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (6)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 4 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Blurred vision (Eye disorders) | 3 (3)
Dry eye (Eye disorders) | 2 (3)
Eye disorders - Other (Eye disorders) | 1 (1)
Floaters (Eye disorders) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 4 (6)
Endocrine disorders - Other (Endocrine disorders) | 2 (3)
Hyperthyroidism (Endocrine disorders) | 2 (4)
Tinnitus (Ear and labyrinth disorders) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Renal calculi (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-03): https://cdn.clinicaltrials.gov/large-docs/66/NCT03663166/Prot_SAP_000.pdf